CLINICAL TRIAL: NCT00278226
Title: Smoking Cessation Among Methadone Maintained Patients
Brief Title: Motivational Program for Smokers Enrolled in a Methadone Maintenance Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Michael Stein, MD, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000452798; R01CA084392 (NIH); RIH-0076-98
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: smoking cessation intervention
Other: educational intervention

SUMMARY:
RATIONALE: Stop-smoking programs may help patients stop smoking and prevent cancer from forming.

PURPOSE: This clinical trial is studying how well a motivational program works in helping smokers enrolled in a methadone maintenance program quit smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of a brief motivational intervention on smoking cessation in smokers enrolled in a methadone maintenance program.

OUTLINE: Patients are assigned to 1 of 2 groups.

* Group 1: Patients undergo assessment at baseline and at 1, 3, and 6 months.
* Group 2: Patients receive a brief motivational intervention at the time of their baseline assessment and undergo assessment as in group 1.

All patients will be offered a 2- to 3-month supply of nicotine patches.

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must be currently enrolled in a methadone maintenance program
* Smokes at least 10 cigarettes a day

PATIENT CHARACTERISTICS:

* Not pregnant
* No concurrent medical condition that precludes the use of nicotine patches

PRIOR CONCURRENT THERAPY:

* No concurrent use of other nicotine replacement therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2001-06; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Nicotine Abstinence | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, MD, Study Chair — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island, United States